CLINICAL TRIAL: NCT03262974
Title: Investigation of the Possible Role of Genetic Polymorphism in Certain Metabolizing Enzymes and Membrane Transporters on Both Plasma Level and Molecular Response of Imatinib in Patients With Chronic Myeloid Leukemia
Brief Title: Effect of Pharmacogenetics on Imatinib Plasma Level and Response
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Sayed Molla, Assistant lecturer, Assiut University
Other Study IDs: Imatinib Pharmacogenetics
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Imatinib; Pharmacogenetics; CML; Plasma level
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from blood samples and frozen at -80 for further analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CML patients with MMR: CYP3A5*3 , CYP2C8*3 , ABCG2 421 C>A and SLC22A1 1222A > G SNPs on the plasma level by HPLC-UV and molecular response of imatinib by PCR
  Interventions: Diagnostic Test: PCR; Diagnostic Test: HPLC-UV
- CML patients without MMR: CYP3A5*3 , CYP2C8*3 , ABCG2 421 C>A and SLC22A1 1222A > G SNPs on the plasma level by HPLC-UV and molecular response of imatinib by PCR
  Interventions: Diagnostic Test: PCR; Diagnostic Test: HPLC-UV

INTERVENTIONS:
Diagnostic Test: PCR — PCR
Diagnostic Test: HPLC-UV — HPLC-UV

SUMMARY:
Imatinib, the tyrosine kinase inhibitor, is used for treatment of Philadelphia positive chronic myeloid leukemia. Despite its efficacy and favorable pharmacokinetic profile, there is a large inter-individual variability in imatinib plasma concentrations, which may lead to treatment failure and disease progression. Polymorphisms in genes related to absorption, distribution, metabolism and excretion of imatinib may affect the bioavailability and consequently the response to the drug.

The study aims to investigate the possible effect of genetic polymorphisms in certain metabolizing enzymes [CYP3A5*3 (rs776746), CYP2C8*3 (rs11572080 and rs10509681)] and membrane transporters [ABCB1 2677G>T/A (rs2032582) and SLC22A1 1222A > G (rs628031)] by PCR on the plasma level (by HPLC-UV) and molecular response (MMR) of imatinib in patients with CML.

The study also aims to provide CML patients with a personalized treatment option, thereby probably improving the response and reducing the side effects.

DETAILED DESCRIPTION:
Introduction:

Chronic myeloid leukaemia (CML) is a myeloproliferative disease with an incidence of one to two cases per 100,000 adults. It accounts for approximately 15% of newly diagnosed cases of leukemia in adults.

The introduction of imatinib, the tyrosine kinase inhibitor (TKI), in the early 21st century is considered a breakthrough in the treatment of CML. In the vast majority of patients, treatment with imatinib induces cytogenetic and even molecular responses with very low or undetectable BCR-ABL1 transcript levels. These patients remain free from progression to blast crisis. However, imatinib does not cure the disease because it is unable to eradicate the leukaemic stem cells, which therefore provides a potential reservoir for relapse.

Despite its efficacy and favorable pharmacokinetic profile, there is a large inter-individual variability in imatinib plasma concentrations, which may lead to treatment failure and disease progression.

Polymorphisms in genes related to absorption, distribution, metabolism and excretion of imatinib may affect the bioavailability and consequently the response to the drug.

Aim of the study:

The study aims to investigate the possible effect of genetic polymorphisms in certain metabolizing enzymes [CYP3A5 * 3 (rs 776746), CYP2C8 * 3 (rs 11572080 and rs 10509681)] and membrane transporters [ABCB1 2677 G>T/A (rs 2032582) and SLC22A1 1222 A > G (rs 628031)] on the plasma level and molecular response (MMR) of imatinib in patients with CML.

These polymorphisms were selected based on their relevance to the pharmacokinetics of imatinib and on their frequency in Caucasians.

The study also aims to provide CML patients with a personalized treatment option, thereby probably improving the response and reducing the side effects.

Patients and methods:

Patients:

The study will include patients with documented hematological, cytogenetic and molecular diagnosis of chronic phase CML, who are on continuous treatment with 400 mg oral dose of imatinib per day for at least 12 month at Medical Oncology Department, South Egypt Cancer Institute (SECI), Assiut. Egypt.

Exclusion criteria are: duration of imatinib therapy less than 12 months, poor compliance to treatment and identification of gene mutation(s) in the kinase domain of BCR- ABL1.

The patients will be divided into 2 groups according to their molecular response to imatinib as follow:

Group I: CML patients with MMR Group II: CML patients without MMR Patients in both groups will be compared as regard the plasma level of imatinib and the selected genetic polymorphisms.

Methods:

Blood sampling:

Three blood samples (3 ml for each) will be collected into EDTA-containing tubes by venipuncture for measurement of imatinib plasma level, measurement of BCR- ABL1 transcription level and for genotyping.

Measurement of Imatinib trough level:

Blood samples will be collected after 24 hours from the previous dose (trough) and after at least 5 days of regular use of the drug to ensure that the steady state is reached. Within 1 hour of collection, the blood samples will be centrifuged at 3,000 rpm for 10 minutes at room temperature and will be stored at -20°C until analysis.

Plasma level of imatinib will be measured by high-performance liquid chromatography with ultraviolet detection (HPLC-UV) according to the method described by Barratt et al.

Measurement of BCR- ABL1 transcription level:

Total RNA will be extracted from peripheral blood leucocytes by the available RNA extraction kits. The BCR- ABL1 transcription level will be quantified by using real-time polymerase chain reaction (PCR) analysis to assess the molecular response to imatinib after 12 months of treatment with imatinib.

Genotyping:

The DNA will be extracted from leukocytes by the available DNA extraction kits and will be stored at -80°C until genotyping.

Genotyping will be performed for CYP3A5 * 3 (rs 776746), CYP2C8 * 3 (rs 11572080 and rs 10509681), ABCB1 2677 G>T/A (rs 2032582) and SLC22A1 1222 A > G (rs 628031) by the PCR

ELIGIBILITY:
Inclusion Criteria:

* Documented hematological, cytogenetic and molecular diagnosis of Philadelphia positive CML
* Imatinib treatment for at least 12 months

Exclusion Criteria:

* Poor compliance to treatment
* identification of gene mutation(s) in the kinase domain of BCR- ABL1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CML patients treated at Medical Oncology Department, South Egypt Cancer Institute (SECI), Assiut. Egypt.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-10-29 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Major molecular response to imatinib | 12 months from starting the drug
  A major molecular response (MMR) to imatinib therapy is defined as a BCR-ABL1 RNA level ≤ 0.1% on the International Scale (a consensus standardized measurement scale intended to allow direct comparison of BCR-ABL1 RNA levels in any laboratory adopting its use). The International Scale was specifically designed so that, by definition, 100% is the median pretreatment baseline level of BCR-ABL1 RNA in early chronic phase CML and a 1,000-fold reduction from baseline is defined as 0.1% (MMR) (Press,

CONTACTS AND LOCATIONS:
Overall Officials: Safwat Mangoura, Study Chair — Pharmacology department, Faculty of Medicine, Assiut University
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Results of genotyping